CLINICAL TRIAL: NCT01833858
Title: The Role of Low Dose HCG in Improving the Quality of Antagonist Protocol in Patient Undergoing ICSI
Brief Title: Human Chorionic Gonadotrophin in an Antagonist Protocol
Acronym: HCG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Elkattan, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol100
Record Dates: First submitted 2013-04-04; First posted 2013-04-17 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo +rFSH (Placebo Comparator): Patients received rFSH injections with a placebo starting on cycle day 3 of the stimulation cycle until the day of hCG trigger administration.
  Interventions: Drug: Placebo
- Low dose HCG with rFSH (Active Comparator): Low dose hCG (200 IU per day) will be given daily with rFSH when at least six follicles of 12 mm will be observed and E2 levels are higher than 600 ng/l, until the day of the hCG trigger administration
  Interventions: Drug: Low dose HCG

INTERVENTIONS:
Drug: Low dose HCG — Low dose hCG (200 IU per day) will be given daily when at least six follicles of 12 mm will be observed and E2 (Estradiol) levels are higher than 600 ng/l, until the day of the HCG trigger administration.
  Other Names: Human chorionic gonadotrophin
  Arms: Low dose HCG with rFSH
Drug: Placebo — Patients received rFSH injections with Placebo starting on cycle day 3 of the stimulation cycle until the day of hCG trigger administration.
  Other Names: saline 0.9%
  Arms: Placebo +rFSH

SUMMARY:
A novel gonadotropin protocol for ovarian stimulation adds low-dose hCG (50- 200 IU) as a source of LH (luteinizing hormone) in the late follicular phase .

This regimen reduces the number of small pre-ovulatory follicles which could reduce the risk of OHSS(ovarian hyper stimulation syndrome). Adequate ovarian hormonal levels , oocyte maturation, avoidance of a premature LH surge, and increased pregnancy rate are the other benefits of this regimen.

HCG might also affect endometrial function, stimulate endometrial growth and maturation and enhance the endometrial angiogenesis. These effects could extend the angiogenesis. These results could lengthen the implantation Window.

Inhibin A is a heterodimer protein and does not begin to increase until just after the increase in oestradiol in the late follicular phase, suggesting secretion by the dominant follicle. Inhibin A secretion is regulated by LH and is associated with paracrine/autocrine action on oocyte maturation. Moreover, it is related to follicular development and size, serving as a marker of follicular maturation after IVF cycles .However, the role of hCG supplementation during COH (controlled ovarian hyperstimulation)is still a matter of debate and more studies is needed. Thus, the objective of this trial was to investigate whether LH activity in the form of low dose hCG in GnRH (Gonadotropin releasing hormone)antagonist cycles would improve the quality of oocytes, level of inhibin A and endometrial vascularity.

DETAILED DESCRIPTION:
* 60 women, where 30 of them will receive low dose HCG with rFSH (group 1), while the other 30 women will receive rFSH (Recombinant Follicle stimulating Hormone) with a placebo (group 2) both using the antagonist protocol as a method of induction in ICSI.
* Women in both groups will be treated with a GnRH antagonist protocol with cetrotide(cetrorelix)
* In Group 1, low dose hCG (200 IU per day) with rFSH will be given daily when at least six follicles of 12 mm will be observed and E2 levels are higher than 600 ng/l, until the day of the hCG trigger administration.
* Group 2 patients received rFSH injections with a placebo starting on cycle day 3 of the stimulation cycle until the day of hCG trigger administration.

In both groups Oocytes will be retrieved 36 h after the hCG trigger shot. All mature eggs retrieved will be fertilized with intracytoplasmic sperm injection (ICSI). Fertilization will be checked at 18 hours post insemination. Embryo quality will be assessed and embryo transfer will occur at day 3.

ELIGIBILITY:
Inclusion Criteria:

1. Indication for ICSI treatment.
2. The presence of one or two functional ovaries.
3. Good responders to ovarian stimulation.
4. The presence of normal uterine cavity
5. Basal (day 2 or 3) serum FSH (follicle stimulating Hormone) levels ≤13 IU
6. No untreated endocrinologic disease

Exclusion Criteria:

1. Abnormal uterine cavity.
2. Basal (day 2 or 3) serum FSH levels ≥13 IU.
3. Poor responders to ovarian stimulation according to the existence of at least two of the following criteria:Advanced maternal age (above 40 years), antral follicles count <5, prior history of poor response to controlled ovarian hyperstimulation (peak E2 <500 pg/ml and/or ≤3 oocytes retrieved).
4. Untreated endocrinologic disease.
5. Azoospermia. all patients should be managed in Cairo,Egypt

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of oocytes | 9 months
Pregnancy rate | 11months

SECONDARY OUTCOMES:
Cost of antagonist treatment | 9 months
Spiral artery Doppler indices | 9 months
  Spiral artery Doppler indices are taken as a marker of subendometrial vascularity.The lowest resistance will be the better vascularity
The percentage of the perifollicular vascularity using power doppler | 9 months
  The percentage of the perifollicular vascularity (<25%,25-50%,%0%-75%,>75%) as a marker of the quality of the oocytes.The more vascularity the better quality

OTHER OUTCOMES:
Serum level of inhibin A | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt